CLINICAL TRIAL: NCT04904783
Title: Low-Dose Radiation Therapy in COVID-19
Brief Title: Low-Dose Radiation Therapy to Lungs in Moderate COVID-19 Pneumonitis: A Case-Control Pilot Study
Acronym: LOCORAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahatma Gandhi Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Niloy Ranjan Datta, Director-Professor & Head, Department of Radiotherapy, Mahatma Gandhi Institute of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGIMS/IEC/RADTHP/215/2021
Record Dates: First submitted 2021-05-25; First posted 2021-05-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: COVID-19; Pneumonia
Keywords: COVID-19; Pneumonia; Low dose radiotherapy; Cytokine storm
MeSH Terms: conditions — COVID-19; Pneumonia; Cytokine Release Syndrome | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: To explore the role of low dose pulmonary radiotherapy (LDRT) in moderate disease category of COVID-19 patients with pneumonitis in terms of the following primary and secondary objectives. The outcome of LDRT in a pilot group of 10 patients (Study group) would be compared with another 10 patients (Control group) who have not given consent for LDRT and/or would not able to be able to lie down still for the entire treatment duration in the radiotherapy unit. This is not a randomized but a case-control study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Active Comparator): 10 patients of confirmed diagnosis of moderate COVID-19 who fulfil the inclusion criteria and give written informed consent would be in study arm. All patients, belong to both study and control groups would receive the same treatment (oxygen support, steroids, anticoagulant therapy, remdesivir and other supportive therapy) as per the Institute guidelines for management of moderate COVID-19 disease. Only low dose radiotherapy would be added to patients in the study arm.
  Interventions: Radiation: Low dose radiotherapy
- Control Arm (No Intervention): 10 patients of confirmed diagnosis of moderate COVID-19 who fulfil the inclusion criteria and have not given written informed consent would be in study arm. These patients would receive the same treatment (oxygen support, steroids, anticoagulant therapy, remdesivir and other supportive therapy) as per the Institute guidelines for management of moderate COVID-19 disease except low dose radiotherapy.

INTERVENTIONS:
Radiation: Low dose radiotherapy — Patients in study group will receive LDRT to both lungs by two parallel opposed fields, antero-posterior (AP) and postero-anterior (PA) to deliver a midplane dose of 0.5 Gy in a single fraction. As this dose is very less, doses to the critical structures including heart and lungs would be very low. All the patients will be treated on Telecobalt unit (Theratronics Phoenix, Canada) and not on the linear accelerator to avoid risks to cancer patients on treatment with linear accelerator. CT based plan will not be undertaken for logistic issues and is also not felt to be mandatory for this LDRT. Dose computation would be carried out by manual dose calculation for the Telecobalt unit.
  Arms: Study arm

SUMMARY:
This pilot case-control study at Mahatma Gandhi Institute of Medical Sciences (MGIMS), Sevagram, India is designed to evaluate the use of low dose radiotherapy (LDRT) in patients with moderate COVID-19 with specific objectives to abrogate the onset of cytokine storm and thus facilitate their early recovery and reduce mortality.

DETAILED DESCRIPTION:
One of the primary attributes to the mortality in coronavirus disease -19 (COVID-19) is acute respiratory distress syndrome (ARDS) induced by severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) mediated cytokine storm (CS).To mitigate the ARDS, an ideal approach would be to diminish the viral load by activating immune cells for CS prevention or to suppress the overactive cytokine-releasing immune cells. The search for ideal pharmaceutical agent/s to take care of SARS-CoV-2 mediated CS is still eluding the clinicians. The only drugs with modest clinical benefit are remdesivir and dexamethasone. The availability of the former is uncertain while an overdependence on steroids could prove counterproductive as evident from increasing incidence of fatal mucormycosis reported in post-COVID patients treated with steroids. The situation for COVID-19 patients successfully treated with steroids is akin to "from frying pan into the fire".

Thus, concerted efforts are needed to prevent the onset of CS in COVID-19. This, would directly help to lower the mortality. One of the approaches being recently investigated worldwide, is the use of single low dose radiotherapy (LDRT) of 0.5 - 1.5 Gy to the lungs before the onset of CS in moderately affected COVID-19 patients requiring oxygen supplementation. This crucial window of opportunity needs to be exploited with LDRT to mitigate the onset of the fatal CS.

LDRT could thus be a potential game changer in the management of COVID-19. LDRT with its multipronged actions may attenuate immune activation and consequently mitigate the production of pro-inflammatory cytokines. A number of centers have reported encouraging outcomes in pilot studies with LDRT. There has been a significant reduction in oxygen requirement within just 72 hours of LDRT, resulting in reduced hospital stay and deaths. This pilot case-control study at MGIMS is designed to evaluate the use of LDRT in patients with moderate COVID-19 with specific objectives to prevent the onset of CS and thus facilitate their early recovery and reduce mortality.

ELIGIBILITY:
Inclusion Criteria:

* Reverse transcription polymerase chain reaction (RT-PCR) / Rapid Ag test positive
* Signed informed consent
* Age ≥ 50 yrs
* Respiratory rate : 25 - 30/min, breathless AND/OR
* Oxygen saturation by pulse oximetry (SpO2) in 90 - 93% on room air (readings taken after 5 mins of stopping oxygen supplementation)
* Rising levels of quantitative-CRP and/or D-Dimer and/or Ferritin in 2 consecutive samples taken 24 hours apart

Exclusion Criteria:

* Patient who have received vaccination for COVID-19 (single / both doses of any approved vaccine)
* Hemodynamic instability in shock and/or systolic BP < 90mm Hg
* Septicemia
* Disseminated intravascular coagulation
* Requiring ventilation
* Unable to lie down supine
* Severe acute respiratory distress with Fraction of inspired oxygen (FiO2) < 100mm Hg
* Cardiac defibrillator/pacemaker in situ
* Lymphocyte count < 1 x 106/ml
* Pregnancy and/or lactating mothers
* HIV and/or HbsAg positive patients

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients dying due to COVID-19 | 28 days from the date of diagnosis
  Compare the number of patients whose death could be ascribed to COVID-19 in the two groups
Mean duration of hospital stay for surviving patients | 28 days from the date of diagnosis / discharge
  Compare the mean duration of hospital stay between the patients surviving in study and control groups

SECONDARY OUTCOMES:
Mean dose of steroid requirement for surviving patients | 28 days from the date of diagnosis
  Compare the mean total dose of steroid required in between the patients surviving in study and control groups
Mean time to completely wean off from Oxygen (02) supplementation for surviving patients | 28 days from the date of diagnosis / discharge
  Compare the mean time to completely wean off from Oxygen supplementation in patients between the patients surviving in study and control groups
Changes in the biochemical profiles of Interleukin-6 (IL-6) | 28 days from the date of diagnosis / discharge
  IL-6 levels in control vs study group patients
Changes in the biochemical profiles of quantitative C reactive protein (CRP) | 28 days from the date of diagnosis / discharge
  Quantitative CRP levels in control vs study group patients
Changes in the biochemical profiles of D-Dimer | 28 days from the date of diagnosis / discharge
  D-Dimer levels in control vs study group patients
Changes in the biochemical profiles of Ferritin | 28 days from the date of diagnosis / discharge
  Ferritin levels in control vs study group patients
Acute pulmonary toxicities that may be attributable to LDRT | 28 days from the date of diagnosis / discharge
  Acute pulmonary toxicities as per the Common Terminology Criteria for Adverse Events (CTCAE) version 5
Total cost of hospital stay following LDRT for surviving patients | 28 days from the date of diagnosis / discharge
  Cost evaluation and comparison between the patients surviving in study and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Niloy R Datta, MD,DNB, Principal Investigator — Dept of Radiotherapy, Mahatma Gandhi Institute of Medical Sciences, India
Locations (2):
- India (2):
  - Mahatma Gandhi Institute of Medical Sciences,, Sevāgrām, Maharashtra
  - Mahatma Gandhi Institute of Medical Sciences, Sevāgrām, Maharashtra

IPD SHARING:
Plan to Share IPD: Yes
Not yet decided. Will decide later after the study results are available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months from date of publication of the final results.
Access Criteria: On request to Principal investigator